CLINICAL TRIAL: NCT00605800
Title: Bone Marrow Derived Adult Liver Stem Cell Recruitment After Major Liver Resections: Correlation With Liver Regeneration and Hepatic Function
Status: Withdrawn | Type: Observational
Why Stopped: Study was closed due to logistical issues.
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Ronald DeMatteo, M.D, Memorial Sloan-Kettering Cancer Center
Other Study IDs: 06-017
Record Dates: First submitted 2008-01-17; First posted 2008-01-31 (Estimated); Last update posted 2009-03-19 (Estimated); Status verified 2009-03

CONDITIONS: Liver Cancer
Keywords: Liver resection
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood

GROUPS / COHORTS (2):
- 1: normal healthy volunteers
  Interventions: Other: blood drawn
- 2: Patients undergoing major liver resections
  Interventions: Other: blood drawn

INTERVENTIONS:
Other: blood drawn — Baseline levels of bone marrow derived liver stem cells from normal healthy volunteers, which will be drawn once Two 5ml blue tubes).
  Groups: 1
Other: blood drawn — At the time of preoperative testing, patients will have two extra test tubes (5cc blue top) of blood drawn for determination of pre-operative base line levels of bone marrow derived liver stem cells in peripheral blood. Intraoperatively, blood will be drawn after liver resection (two tubes of 5cc blue top). Two extra tube of blood will be drawn at the same time of routine postoperative blood drawing to determine levels of bone marrow derived liver stem cells in peripheral blood on post-operative days #1, and #3.
  Groups: 2

SUMMARY:
The results of this study may or may not establish useful baseline data, which will help us understand how bone marrow derived adult liver stem cells behave in normal healthy adults/volunteers (the control group), and in patients undergoing liver surgery. The bone marrow is located within your bones and is the organ which is responsible to produce blood cells and stem cells. Bone marrow derived adult liver stem cells are normal cells in your bone marrow. These liver stem cells have the capacity to regenerate or in other words to rebuild the liver after liver surgery, a process called liver regeneration. These cells are very important for the liver to regrow its tissue after liver surgery. These cells are thought to be activated in times of need by the liver.

Situations like liver surgery are one of these occasions when the liver will need the "extra help" from these stem cells.

The results of this study will establish the baseline data necessary for the understanding of how to harness the ability of these stem cells in times of liver surgery. Improvements in the ability of the liver to regrow after surgery is thought to decrease complications related to liver surgery. Harnessing this unique ability of stem cells may be utilized in the future to enhance the regrowing process of liver tissue after liver surgery, called liver regeneration.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ or equal to 18 years old).
* Patients scheduled for resection of 3 or more liver segments for any indication, with or without other planned procedures.

Or

* Normal healthy volunteers (control).

Exclusion Criteria:

* Chemotherapy or GCSF treatment in the preceding 4 weeks.
* CHILD'S classification B or above.
* Presence of active infection.
* History of lymphoma or leukemia.
* Normal healthy volunteers who underwent chemotherapy treatment at any stage of their life will be excluded.
* Normal healthy volunteers who are under any active treatment for any active illness will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: MSKCC clinics Normal healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-03; Primary Completion 2009-03 (Estimated); Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
To determine qualitatively and quantitatively whether bone marrow derived liver associated stem cells are mobilized from the bone marrow in patients undergoing major liver resections (3 or more liver segments). | conclusion of study

SECONDARY OUTCOMES:
To determine whether a difference exist in the baseline levels of bone marrow derived liver associated stem cells between normal healthy subjects/ volunteers and cancer patients prior to liver surgery. | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Ronald DeMatteo, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org